CLINICAL TRIAL: NCT04803955
Title: Efficacy and Safety of Kukoamine B Mesilate in Sepsis Patients: a Multicentre, Randomised, Double-blind, Placebo-controlled, Phase 2 Trial
Brief Title: Efficacy and Safety of Kukoamine B Mesilate in Sepsis Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Chasesun Pharmaceutical Co., LTD (Industry)
Collaborators: Southwest Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-KB201
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 16mg,KB (Experimental): Group A:16mg,Q8h±3min,Day1-Day7
  Interventions: Drug: 16mg，KB
- Placebos (Placebo Comparator): Group B:Placebos,Q8h±3min,Day1-Day7
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 16mg，KB — 16mg,Q8h±3min,Day1-Day7
  Arms: 16mg,KB
Drug: Placebos — 16mg,Q8h±3min,Day1-Day7
  Arms: Placebos

SUMMARY:
Phase II study of Kukoamine B Mesilate in Sepsis Patients

DETAILED DESCRIPTION:
To Assess Efficacy,Safety,Pharmacokinetics of Kukoamine B Mesilate in Sepsis Patients

ELIGIBILITY:
Inclusion Criteria:

* (1) The age of ≥ 18 years of age and ≤ 85 years of age, gender is not limited;
* (2) Meeting the diagnostic criteria for sepsis 3.0, i.e. sequential organ failure score (SOFA) increased by ≥2 points from baseline for patients with confirmed or suspected infection;
* (3) Confirmed or suspected bacterial infection (Pulmonary, abdominal，urinary system or hematogenous infections);
* (4) Infection-related organ failure does not exceed 48 hours; organ failure is defined as circulation, (SOFA) ≥ 3 points in at least one organ or system of the respiratory, kidney, liver, coagulation and central nervous system;
* (5) Childbearing age within six months without child care plan and agreed to take effective measures during the study of contraception;
* (6) Patients or guardians signed informed consent.

Exclusion Criteria:

* (1) Pregnancy or lactation women；
* (2) Patients are expected to live less than 48 hours;
* (3) Patients had poor control of malignant tumor, end-stage lung disease and other end-stage diseases, or had acardiac arrest，acute pulmonary embolism，blood transfusion response and acute coronary syndrome within 4 weeks prior to enrollment;
* (4) The patient has the following chronic organ dysfunction or immunosuppression (based on the chronic health scoring assessment of the APACHE II score) : 1) heart: New York heart association cardiac function IV; 2) breathing: chronic obstructive, obstructive, or vascular lung disease can lead to severe restrictions on activities, i.e. the inability to go upstairs or to do housework; Or clear chronic hypoxia, CO2 retention, secondary real erythrocyte, severe pulmonary hypertension (mPAP> 40 mmHg) or respiratory muscle dependence; 3) kidneys: receiving long-term dialysis; 4) liver: liver cirrhosis confirmed by biopsy and clear portal hypertension; The upper digestive tract hemorrhage caused by portal hypertension; Or previous liver failure/hepatic encephalopathy/hepatic coma; 5) of immune function: accept the treatment of impact resistance to infection, such as immune suppression therapy, chemotherapy, radiotherapy or chemotherapy within 6 months, long-term (continuous use ≥3 weeks) use of glucocorticoids or recent (within 5 days before screening) cumulative use of prednisone or equivalent dose ≥100mg , or sickness impact resistance to infection, such as leukemia, lymphoma and AIDS);
* (5) Previous solid organ or bone marrow transplantation;
* (6) Plant survival status;
* (7) Confirmed or highly suspected of acute infectious diseases such as viral hepatitis activity , or clinically confirmed active tuberculosis;
* (8) Patients with sinus bradycardia (less than 60 per minute);
* (9) Uncontrolled bleeding in the past 24 hours（Clinical judgment requires transfusion support）;
* (10) Large area burns or chemical burns (III degree burns area > 30% BSA);
* (11) The average arterial pressure was < 65 mmHg after adequate liquid resuscitation and vasoactive drug therapy;
* (12) Acute myeloid hematopoiesis was characterized by a lack of severe granulocytes (ANC < 500 / mm3);
* (13) Allergic to the active ingredient or its auxiliary materials;
* (14) The medication patients are using may severely affect the metabolism of the drug;
* (15) Patients and (or) guardians have signed a Do Not Rescue (DNR), or decided to withdraw life support (withdraw) or restrict life support for the intensity (withhold) and sign the informed consent form;
* (16) Participated in clinical intervention test in 3 months;
* (17) The subject is a researcher or his immediate family member, or may have improper informed consent;
* (18) The investigator considers it inappropriate for the patient to participate in this test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Delta SOFA (ΔSOFA) | Day 8 after the first dose (Within 24 hours after the last dose on day 7)
  Change in SOFA scale from baseline.

SECONDARY OUTCOMES:
Clinical Outcome Composite Endpoint | 28 days after the first dose
  Proportion of patients with 28-day all-cause deaths and continuing ICU stay after the first dose.
Proportion of patients with 7-day all-cause deaths | 7 days after the first dose
  Proportion of patients with 7-day all-cause deaths after first dose.
Proportion of patients transferred out of ICU | 7 days after the first dose
  Proportion of patients transferred out of ICU within 7 days after first dose.
Quantification of IL-6 | Day 2, 4 , 8 after the first dose (Within 24 hours after the last dose on day 7)
  Change of IL-6 from baseline on day 2,4,8 after first dose (Within 24 hours after the last dose on day 7).
Delta SOFA (ΔSOFA) | Day 1, 3, 5 after the first dose
  Change in SOFA scale from baseline on day 1,3 ,5 after first dose.
Duration of use and abstention of life support treatment | 28 days after the first dose
  Duration of use and abstention of life support treatment (vasoactive drugs, mechanical ventilation, CRRT) .
Duration of ICU stay and absence | 28 days after the first dose
  Duration of ICU stay and absence within 28 days after the first dose.
Rate of adverse events/serious adverse events | From date of singing informed consent until the 29 days after the first dose
  Observe all the participants in any adverse events occurred during the period of clinical research, including clinical symptoms and signs of life, an abnormal in laboratory tests, record its clinical characteristics, severity, occurrence time, duration, treatment and prognosis, and determine its and the correlation between test drugs. CTCAE v5.0 standard was used to evaluate drug safety.

OTHER OUTCOMES:
Area under the curve at steady state (AUCss) | Day 1 and Day 7
  determination of area under curve
Peak plasma concentration at steady state (Cmaxss) | Day 1 and Day 7
  determination of Cmax
Trough plasma concentration at steady state (Cminss) | Day 1 and Day 7
  determination of Cmin
Correlation between the exposure of Kukoamine B Mesilate and its efficacy | Day 8 after the first dose (Within 24 hours after the last dose on day 7)
  Correlation between the exposure of Kukoamine B Mesilate and change in SOFA scale from baseline.
Correlation between the exposure of Kukoamine B Mesilate and hepatic-related treatment-related adverse events | Day 1 to Day 8
  Correlation between the exposure of Kukoamine B Mesilate and hepatic-related treatment-related adverse events of interest as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided